CLINICAL TRIAL: NCT00444756
Title: Jet Injection of 1% Buffered Lidocaine Versus Topical ELA-Max for Anesthesia Prior to Peripheral Intravenous Catheterization in Children
Brief Title: Jet Injection of 1% Buffered Lidocaine Versus Topical ELA-Max for Anesthesia Prior to Intravenous (IV) Catheterization in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norton Healthcare (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 622.04
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2007-03

CONDITIONS: Pain
Keywords: local anesthesia; analgesia; peripheral IV; Local anesthesia prior to peripheral IV insertion
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: J-tip jet injection of 1% buffered lidocaine

SUMMARY:
This trial is a comparison of the anesthetic effectiveness of J-Tip needle-free jet injection of 1% buffered lidocaine to the anesthetic effectiveness of topical 4% ELA-Max for peripheral intravenous catheter (PIV) insertion. The researchers hypothesize that the jet injection of lidocaine will provide superior anesthesia to the ELA-Max prior to PIV insertion.

DETAILED DESCRIPTION:
A prospective, block-randomized, controlled trial comparing J-Tip jet injection of 1% buffered lidocaine to a 30-minute application of 4% ELA-Max for topical anesthesia in children 8-15 years old presenting to a tertiary care pediatric emergency department for PIV insertion. All subjects recorded self-reported Visual Analogue Scale (VAS) scores for pain at time of enrollment and pain of PIV insertion. Jet injection subjects also recorded pain of jet injection. Subjects were videotaped during jet injection and PIV insertion. Videotapes were reviewed by a single blinded reviewer for observer-reported VAS pain scores for jet injection and PIV insertion.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8-15 years requiring a PIV as part of their management in the emergency department.

Exclusion Criteria:

* Excluded from the study if they reported use of analgesic medication within 6 hours of enrollment,
* Had a Glasgow Coma Score < 15,
* A baseline screening VAS pain score > 20 mm, or
* A history of skin hypersensitivity or lidocaine allergy,
* Were incapable of self-reporting a pain score,
* Had a known neurological condition that alters pain perception,
* Had methemoglobinemia, or
* Did not speak or understand English.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70
Dates: Start 2005-04; Study Completion 2006-04

PRIMARY OUTCOMES:
VAS pain scores for the PIV insertion as judged by the patients and the blinded observer.

SECONDARY OUTCOMES:
Secondary outcome measures included patient and blinded observer VAS scores for pain of jet injection, patient and blinded observer scores for anxiety of PIV insertion, nursing satisfaction of placing the PIV with jet injection or ELA-Maxâ, nursing diffi

CONTACTS AND LOCATIONS:
Overall Officials: In K Kim, MD, Study Director — Department of Pediatric Emergency Medicine, Department of Pediatrics, Kosair Children's Hospital, University of Louisville, Louisville, Kentucky
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Spanos S, Booth R, Koenig H, Sikes K, Gracely E, Kim IK. Jet Injection of 1% buffered lidocaine versus topical ELA-Max for anesthesia before peripheral intravenous catheterization in children: a randomized controlled trial. Pediatr Emerg Care. 2008 Aug;24(8):511-5. doi: 10.1097/PEC.0b013e31816a8d5b. PMID 18645542